CLINICAL TRIAL: NCT01499966
Title: Assessment of Tubigrip Versus Plaster of Paris in the Treatment of Grade 1 and 2 Lateral Ankle Sprains
Brief Title: Comparison of Plaster of Paris Against Tubigrip for the Treatment of Lateral Ankle Sprains
Acronym: POPTuLAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liaquat National Hospital & Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRahimnajjad
Record Dates: First submitted 2011-10-31; First posted 2011-12-26 (Estimated); Last update posted 2011-12-26 (Estimated); Status verified 2011-12

CONDITIONS: Ankle Injuries
Keywords: Lateral Ankle Sprain; Plaster of Paris; Tubigrip
MeSH Terms: conditions — Ankle Injuries | interventions — Calcium Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- group POP (Experimental): PLASTER OF PARIS
  Interventions: Procedure: Plaster of Paris/ Tubigrip
- TG (Experimental): TUBIGRIP
  Interventions: Procedure: Plaster of Paris/ Tubigrip

INTERVENTIONS:
Procedure: Plaster of Paris/ Tubigrip — After informed consent was obtained the patients were randomized such that each patient was allocated to use either a Tubigrip (Group A) or Plaster of Paris (Group B). The standardized treatment in the form of RICE (Rest, Ice, Compression and Elevation) protocol was given to all patients. The Patients were randomized using the Block randomization. One hundred and twenty six white papers were taken and "TG" for Tubigrip and "POP" for Plaster of Paris were written and the patients were allowed to pick the envelope of their choice. The authors were blinded till the opening of the envelope by the patients. Patient's usage of analgesia in form of Paracetamol was specifically noted. The patients in TG group receive the Tubigrip treatment and the patients in POP group were given a below knee plaster cast. Patients were instructed to follow up at 2 weeks and then at 6 weeks

SUMMARY:
Until now very few studies have been done to compare the efficacy of tubigrips or plaster of paris in the treatment of lateral ankle sprains, the investigators aim to compare the tubigrip against plaster of paris in the treatment of lateral ankle sprains.

DETAILED DESCRIPTION:
200 patients were enrolled after meeting inclusion criteria.All patients gave the verbal as well as written consent for inclusion in the study. The hospital committee ethical review board gave the permission for this study. Only 126 patients agreed to participate in the study. After informed consent was obtained the patients were randomized such that each patient was allocated to use either a Tubigrip (Group A) or Plaster of Paris (Group B)using the Block randomization. The patients in TG group receive the Tubigrip treatment and the patients in POP group were given a below knee plaster cast. Patients were instructed to follow up at 2 weeks and then at 6 weeks. The functional score and pain were used as outcomes of the study

ELIGIBILITY:
Inclusion Criteria:

* age 18-40 years
* grade 1 and 2 ankle sprains
* permanent residents in place of study
* no concomitant bone pathology
* have not been recruited in other trial simultaneously

Exclusion Criteria:

* Patients with age <18 years
* injury >48 hours, fractures
* multiple injuries
* any neurological or musculoskeletal illness
* any co-morbid associated with long term disabilities
* grade 3 lateral ankle sprains

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2011-01; Primary Completion 2011-07 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
pain, karlsson score | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Zaki Idrees, FRCS, Study Chair — Liaquat National Hospital
Locations (1):
- Liaquat National Hospital, Karachi, Sindh, Pakistan

REFERENCES:
- [Derived] Naeem M, Rahimnajjad MK, Rahimnajjad NA, Idrees Z, Shah GA, Abbas G. Assessment of functional treatment versus plaster of Paris in the treatment of grade 1 and 2 lateral ankle sprains. J Orthop Traumatol. 2015 Mar;16(1):41-6. doi: 10.1007/s10195-014-0289-8. Epub 2014 Mar 27. PMID 24671488